CLINICAL TRIAL: NCT02725190
Title: Effects of Sleep Deprivation on Diaphragm Command During an Inspiratory Endurance Trial in Healthy Volunteers.
Acronym: NoSleepDiaph
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: NoSleepDiaph
Record Dates: First submitted 2016-03-25; First posted 2016-03-31 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Sleep Deprivation; Healthy Volunteers; Diaphragm
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Other): Normal sleep night.
  Interventions: Behavioral: Normal sleep night
- Group 2 (Other): Sleepless night.
  Interventions: Behavioral: Sleepless night

INTERVENTIONS:
Behavioral: Sleepless night — Each subject will undergo 28 hours of sleep deprivation.
  Arms: Group 2
Behavioral: Normal sleep night — Normal sleep at home before trial.
  Arms: Group 1

SUMMARY:
The purpose of this study is to assess the impact of sleep deprivation on subjective inspiratory endurance in healthy subjects.

DETAILED DESCRIPTION:
Sleep in intensive care unit is altered and few studies have suggested that sleep deprivation (SD) could impact respiratory muscle endurance. A lack of inspiratory endurance could lengthen weaning from invasive ventilation. The purpose of this study is to confirm whether SD alters inspiratory endurance and to identify brain mechanisms involved in SD-induced decreased endurance. A group of 20 male healthy subjects will perform an inspiratory load trial after a normal sleep night and after a sleepless night. Electrophysiological parameters (EEG, motor evoked potentials) of the inspiratory motor command and sensory perceptions will be assessed before, during and after each trial.

ELIGIBILITY:
Inclusion Criteria:

* Male adult volunteers
* Aged 25 to 45 years
* Regularly sleeping more than 6 hours per night
* Not excessive coffee consumers (< 3 expressos / day)
* Non smokers
* Absence of respiratory, cardiac, muscular or neurological disease or diabetes
* With a neutral Horne & Ostberg score

Exclusion Criteria:

* Previous history of respiratory disease or otorhinolaryngological (asthma, respiratory allergies, swallowing disorders, oropharyngeal malformations)
* History of epilepsy or syncope during sleep deprivation
* Taking medications that interfere with sleep (antidepressants, benzodiazepines…)

Ages: 25 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-04; Primary Completion 2017-08 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Time, in minutes, measured from the beginning of the inspiratory endurance test and the end, defined by the patient's wish to stop. | The day after one normal night or one sleepless night.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Drouot, MD, PhD, Principal Investigator — CHU Poitiers
Locations (1):
- CHU de Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Westphal WP, Rault C, Robert R, Ragot S, Neau JP, Fernagut PO, Drouot X. Sleep deprivation reduces vagal tone during an inspiratory endurance task in humans. Sleep. 2021 Oct 11;44(10):zsab105. doi: 10.1093/sleep/zsab105. PMID 33895822